CLINICAL TRIAL: NCT05344339
Title: Billroth-II Modified and Roux-en-Y Reconstruction After Distal Gastrectomy for Gastric Cancer: an Open-label Randomized Control Trial
Brief Title: Billroth-II Modified Versus Roux-en-Y After Distal Gastrectomy for Gastric Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15/GCN-HDDD
Record Dates: First submitted 2022-04-08; First posted 2022-04-25 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2023-12

CONDITIONS: Gastric Cancer; Distal Gastrectomy
Keywords: Gastric Cancer; Distal gastrectomy; Reconstruction; Gastric adenocarcinoma; Roux-en-Y
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gastroenterostomy

STUDY DESIGN:
Intervention Model Description: Open label randomized control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Billroth-II modified (Experimental): An opening will be made at jejunum 25 cm from Treitz's ligament. Another at greater curvature of the stomach right above transected line. A straight stapling device will be used to make isoperistaltic anastomosis at posterior wall of the stomach. After checking for bleeding, common entry hole will be closed using running suture and 3 -5 sutures to attach afferent loop to the remnant stomach
  Interventions: Procedure: Distal gastrectomy
- Roux-en-Y (Active Comparator): Jejunum will be transected 25 to 30 cm from Treitz's ligament. Marginal vessels will be transected if needed to make sure the loop will reach the stomach without tension. Isoperistaltic gastrojejunostomy will be made at posterior wall of the stomach. After checking for bleeding, common entry hole will be closed using running suture. Jejunojejunal mesenteric defect and Petersen's defect will be closed.
  Interventions: Procedure: Distal gastrectomy

INTERVENTIONS:
Procedure: Distal gastrectomy — Reconstruction after Distal Gastrectomy

SUMMARY:
There are Billroth-I, Billroth-II, Billroth-II with Braun, and Roux-en-Y reconstruction after distal gastrectomy.

Hypothesis: Billroth-II modified method is non-inferior to Roux-en-Y method in terms of reducing reflux esophagitis after distal gastrectomy for gastric cancer patients.

DETAILED DESCRIPTION:
Since the first gastrectomy by Theodore Billroth in 1881, this procedure remained a curative treatment for gastric cancer. Reconstruction method after gastrectomy may affect complication rates, post-operative nutritional status, and quality of life (QoL). There are several reconstruction methods for distal gastrectomy, including Billroth I (B-I), Billroth II (B-II), Roux-en-Y (R-Y). B-I and B-II were considered better than R-Y in terms of shorten operation time and lessen blood loss due to technical simplicity. In contrast, R-Y was better in terms of preventing bile reflux and remnant gastritis, which can increase remnant stomach cancer and worsen QoL. However, long term QoL was similar between B-I and R-Y in some randomized controlled trials. Although bile reflux was higher in B-I and B-II groups, remnant gastric cancer was similar between 3 groups in this study. In brief, which one is the ideal reconstruction after distal gastrectomy is still controversial.

At our center, reconstruction after distal and sub-total gastrectomy including B-I, B-II, B-II with Braun anastomosis, and R-Y, depended mostly on surgeons' preferences. From 2018, to decrease bile reflux rate while not increasing operation time, we applied modified B-II technique with 3-5 sutures between the afferent loop to the gastric remnant. This study was conducted to evaluate the efficacy of this method by comparing it with the R-Y method.

ELIGIBILITY:
Inclusion Criteria:

* Patients confirmed with gastric cancer
* Indicated for radical distal gastrectomy (cT1 to cT4a, any N, M0; according to AJCC/UICC 8th TNM staging for gastric cancer)
* Age from 18- to 80-year-old
* Agreed to participate in study with written inform consent

Exclusion Criteria:

* Pregnant patients
* An American Society of Anesthesiology (ASA) score of higher than 4
* Concurrent cancer or history of previous other cancers
* Previous gastrectomy
* Complications including bleeding, perforation required emergency gastrectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2022-10-08 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Reflux esophagistis | on the 12th month after surgery
  Findings of reflux esophagitis according to Los Angeles classification via endoscopy

SECONDARY OUTCOMES:
Early complications | 30 days after surgery
  Rate of any complications happened intraoperative and 30-days post-operative
Operative time | Intraoperative
  Time from first incision to finishing abdomen closure, measured by surgical nurse
Time for making anastomosis | Intraoperative
  Time from jejunal stapler opening (for B-II) or from jejunal separating (for R-II) to finishing enhancing suture (including duodenal stump enhancement)
Blood loss | Intraoperative
  Weighing of sucked blood and gauze, minus weighing of dry gauze
Length of post-operative hospital stay | 30 days after surgery or until mortality
  Number of days from date of surgery until date of discharge or mortality
Post gastrectomy syndromes | from 30 days to 1 years after surgery
  Rate of post gastrectomy syndromes after gastrectomy
Bodyweight | on the 3rd, 6th, and 12th month after surgery
  Changing of patient's weight at the follow-up time compare to weight before surgery
Serum total protein | on the 3rd, 6th, and 12th month after surgery
  Changing of patient's serum total protein at the follow-up time compare to serum protein before surgery
Serum albumin | on the 3rd, 6th, and 12th month after surgery
  Changing of patient's serum albumin at the follow-up time compare to serum albumin before surgery
Hemoglobin | on the 3rd, 6th, and 12th month after surgery
  Changing of patient's hemoglobin at the follow-up time compare to hemoglobin before surgery
Changing of Gastric remnant gastritis | on the 6th, and 12th month after surgery
  Grade of gastric remnant gastritis according to RGB classification (for endoscopy) and updated Sydney classification (for histology)
Changing of Residual food | on the 6th, and 12th month after surgery
  Grade of Residual food according to RGB classification via endoscopy
Changing of bile reflux | on the 6th, and 12th month after surgery
  Finding of bile reflux according to RGB classification via endoscopy
Changing of GSRS score | on the 3rd, 6th, and 12th month after surgery
  Patient's quality of life evaluated using the Gastrointestinal Symptom Rating Scale (GSRS) questionnaire
6th month reflux esophagistis | on the 6th month after surgery
  Findings of reflux esophagitis according to Los Angeles classification via endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Long D Vo, MD, PhD, Principal Investigator — University Medical Center HCMC, VN
Locations (1):
- University Medical Center Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No